CLINICAL TRIAL: NCT04289636
Title: Comparison of Two Approaches for Improving Long-term Weight Loss Among Individuals With Severe Obesity
Brief Title: Self-compassion and Nutrition (SCAN) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Jessica Unick, Assistant Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1569066
Record Dates: First submitted 2020-02-27; First posted 2020-02-28 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Obesity; Weight Loss
Keywords: self-compassion; exercise; nutrition; physical activity
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight loss and self-compassion (Experimental): Participants will receive a 15-week behavioral weight loss program which teaches strategies for changing diet and exercise behaviors. This will consist of a combination of group and individual sessions. Group classes will be delivered remotely via a video-conferencing platform. This will be followed by an 8-week mindfulness-based self-compassion program which combines the skills of mindfulness and self-compassion as a means for improving emotional resilience, well-being, and weight control.
  Interventions: Behavioral: Behavioral weight loss program; Behavioral: Self-compassion
- Weight loss and nutrition/cooking education (Active Comparator): Participants will receive a 15-week behavioral weight loss program which teaches strategies for changing diet and exercise behaviors. This will consist of a combination of group and individual sessions. Group classes will be delivered remotely via a video-conferencing platform. This will be followed by an 8-week nutrition and cooking education program which will provide basic nutrition knowledge and cooking skills for healthy eating.
  Interventions: Behavioral: Behavioral weight loss program; Behavioral: Nutrition and cooking education

INTERVENTIONS:
Behavioral: Behavioral weight loss program — Using a combination of individual (~1x/month) and group-based (~3x/month) meetings, participants will be taught behavioral approaches for changing diet and exercise behaviors. This intervention will be 15 weeks in duration and will be delivered remotely using a video-conferencing platform.
Behavioral: Self-compassion — This 8-week, group-based program will help train individuals on how to handle difficult emotions with greater ease, how to transform difficult relationships, and how to motivate and encourage oneself, rather than being self-critical.
  Arms: Weight loss and self-compassion
Behavioral: Nutrition and cooking education — This 8-week, group-based program will help individuals to improve the quality of their diet through nutrition education and basic cooking skills for preparing healthy meals.
  Arms: Weight loss and nutrition/cooking education

SUMMARY:
The purpose of this study is to examine the feasibility of two approaches for improving long-term weight loss success among individuals with severe obesity. All participants will receive a 15-week, standard behavioral weight loss program followed by either 8 weeks of a mindfulness self-compassion intervention or 8 weeks of a nutrition and cooking education intervention (determined via randomization procedures). Assessments of weight, physical activity, and other weight-related and psychosocial factors will occur at baseline, 4 months, 6 months, and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* BMI between 40 - 55 kg/m2
* Female
* Score high on internalized weight bias

Exclusion Criteria:

* Presence of any condition that would limit one's ability to exercise (i.e., orthopedic limitations)
* Recent weight loss (≥15 pounds within the past 6 months)
* History of bariatric surgery
* Current or recent enrollment (completed <1 year ago) in a weight loss program at the Weight Control and Diabetes Research Center
* Currently taking any weight loss or other medication that could alter one's metabolism
* Women who are pregnant, planning on becoming pregnant in the next 6 months, or those pregnant within the past 6 months
* Serious psychiatric disorder (e.g., psychosis, major depression, suicidality) -
* Participants with a history of diabetes or heart disease will be considered for this study only if their heart disease or diabetes is well controlled, and physician consent will be required.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Recruitment feasibility will be assessed by the number of participants screened and enrolled | At the end of the study, up to 9 months post-baseline
  Recruitment feasibility will be assessed by the number of participants screened and enrolled
Session attendance will be assessed by calculating the overall session attendance (# of sessions completed/# of sessions possible). | 6 months
  The feasibility of the intervention will be assessed by calculating the overall session attendance
Acceptability of the intervention (retention) will be determined by the percentage of participants completing the 9-month assessment visit | 9 months
  Acceptability of the intervention (retention) will be determined by the percentage of participants completing the 9-month assessment visit

SECONDARY OUTCOMES:
Percent weight change at 6 months | 6 months after study enrollment
Percent weight change at 9 months | 9 months after study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Unick, PhD, Principal Investigator — The Miriam Hospital's Weight Control & Diabetes Research Center
Locations (1):
- The Miriam Hospital's Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided